CLINICAL TRIAL: NCT03891381
Title: Electromyographic Monitoring and Postoperative Recovery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution
Sponsor: Endeavor Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EH13-032
Record Dates: First submitted 2019-03-25; First posted 2019-03-27 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2020-02

CONDITIONS: Postoperative Residual Neuromuscular Blockade

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to a qualitative (peripheral nerve stimulator) or quantitative (Tetragraph) monitor
Who Masked: Participant
Masking Description: Patients will be under anesthesia and unaware of type of monitoring used in the operating room
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Tetragraph (Experimental): Patients will be randomized to receive quantitative monitoring in the operating room. Neuromuscular management will be guided by information provided by the monitor
  Interventions: Device: Tetragraph quantitative monitoring
- Qualitative monitoring (Active Comparator): The screen of the Tetragraph will be covered so that information is not provided to the clinician. The monitor will therefore function as a standard peripheral nerve monitor (clinicians will only observe the response to nerve stimulation)
  Interventions: Device: Tetragraph quantitative monitoring

INTERVENTIONS:
Device: Tetragraph quantitative monitoring — Neuromuscular monitoring will be guided by information provided by the Tetragraph

SUMMARY:
Residual neuromuscular blockade (weakness) is a common occurrence in the postanesthesia care unit when muscle relaxant drugs have been used in the operating room. The only method of reliably detecting residual neuromuscular blockade is through the use of quantitative neuromuscular monitors. These devices measure and quantify the degree of muscle weakness and display the results on a screen. When using train-of-four (TOF) nerve stimulation, the ratio of the fourth muscle contraction (twitch) to the first twitch will be displayed; when this ratio is 90% (or 0.9) or greater, full recovery of muscle strength is present, and the endotracheal tube can be safely removed. At the present time, there is only one commercially available quantitative monitor produced in the United States -the TOF-Watch. The TOF-Watch is not used by many clinicians because it requires experience to obtain accurate results, is expensive, and is subject to interference by factors in the operating room. The aim of this investigation is to examine a new quantitative monitor (the TetraGraph, an electromyography (EMG) device) in the clinical setting. Patients will be randomized to receive either electromyography monitoring (EMG group-using the TetraGraph) or qualitative peripheral nerve stimulator monitoring (PNS group-the standard type of neuromuscular monitoring used at NorthShore University HealthSystem). The primary endpoint of the investigation is the incidence of postoperative residual blockade (defined as a TOF ratio < 0.9 with TOF-Watch, the current "gold standard quantitative monitor). Secondary endpoints include a variety of standard clinical recovery variables.

DETAILED DESCRIPTION:
Although anesthesiologists recognize that residual neuromuscular block can adversely affect postoperative recovery, a high percentage of patients continue to arrive in the PACU with TOF ratios < 0.9. An important reason this problem occurs is that anesthesiologists rarely use quantitative neuromuscular monitoring in the operating room. In current anesthesia practices, clinicians typically use standard peripheral nerve stimulators (qualitative neuromuscular monitors) and / or clinical tests of muscle strength to detect residual muscle weakness at the end of surgical procedures. Qualitative nerve stimulators/monitors are routinely used in the operating rooms; TOF electrical stimuli are applied to a peripheral nerve, and the contractions of the innervated muscle observed. However, visual or tactile assessment of TOF stimulation using these monitors is only effective in detecting profound levels of muscle weakness (TOF ratios < 0.4) Therefore, qualitative nerve stimulators are unable to reliably detect clinically relevant neuromuscular block (TOF ratios of 0.5-0.9). Clinical assessment of patients for signs of muscle weakness (head-lift, hand squeeze) is also an insensitive method of detecting residual neuromuscular block, since many patients can perform these tests with TOF ratios as low as 0.5.

In order for clinicians to reliably exclude residual neuromuscular blockade, quantitative neuromuscular monitoring should be used. At the present time, only one stand-alone quantitative monitor has been produced for clinical use, the TOF-Watch (Blue Star Enterprises, Chanhassen, Minnesota-no longer manufactured). This technology (acceleromyography (AMG)) uses a piezoelectric crystal to sense the acceleration of muscle contractions, and converts this data into a displayed TOF ratio (0-100%). Although the use of the TOF-Watch has been demonstrated to reduce the risk of residual blockade, the routine application of this monitor by clinicians has been limited by a number of factors, related to complexity of use in the operating room.. There is an urgent need for an easy-to-use and accurate quantitative neuromuscular monitor in the clinical setting. Recently, a new device has been developed that uses electromyography (EMG) technology to assess recovery of muscle function in the clinical setting (the TetraGraph). This EMG device measures electrical activity (compound muscle action potentials) following nerve stimulation (usually at the thenar eminence after ulnar or median nerve stimulation). When TOF stimuli are provided, this data is then converted to a measurable TOF ratio (from 0-1.0 or 0-100%). In a study completed at NorthShore University HealthSystem, the investigators compared the applicability (ease of use, equipment need, etc.), repeatability (precision or internal consistency), and performance (agreement with established standard, bias) of this EMG technology to the TOF-Watch (the current clinical "gold standard" quantitative neuromuscular monitor). The subsequent analysis suggested that EMG monitoring accurately measures onset and recovery of neuromuscular function in the operating room.

The use of quantitative neuromuscular monitoring in the operating room should allow for more rational management of dosing and reversal of NMBAs. Furthermore, if incomplete neuromuscular recovery is detected at the end of a surgical procedure, tracheal extubation can be delayed until full recovery of muscle strength has occurred. Therefore, fewer patients should leave the operating room with muscle weakness, and the risks/complications of residual blockade in the PACU reduced. The aim of this clinical investigation is to determine whether EMG monitoring in the operating room reduces the incidence of postoperative residual blockade (measured at the time of tracheal extubation and on arrival to the PACU). During the PACU admission, patients will also be assessed for potential complications related to incomplete neuromuscular recovery (signs and symptoms of muscle weakness, episodes of hypoxemia and airway obstruction, prolonged PACU length of stay). Patients will be randomized to receive either electromyography monitoring (EMG group-TetraGraph) or qualitative peripheral nerve stimulator monitoring (PNS group) in the operating room. The primary endpoint is the incidence of postoperative residual block (defined as a TOF ratio < 0.9 with the TOF-Watch monitor). Secondary endpoints include a variety of clinical recovery variables listed below.

ELIGIBILITY:
Inclusion Criteria: American Society of Anesthesiologists Status I - III patients undergoing surgery requiring neuromuscular blockade

-

Exclusion Criteria:

presence of an underlying neuromuscular disease; use of drugs known to interfere with neuromuscular transmission (antiseizure medications, anticholinesterases, magnesium sulfate); renal insufficiency (serum creatinine > 1.8 mg/dL) or renal failure.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-10-20 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative residual neuromuscular blockade | 15 minutes
  the percentage of patients admitted to the postanesthesia care unit with train-of-four ratios < 0.9 will be determined

SECONDARY OUTCOMES:
Incidence of hypoxemic events in the postanesthesia care unit | 60 minutes
  The number of patients with episodes of oxygen saturations < 95% will be determined
Airway obstruction | 60 minutes
  the number of episodes of clinically-observed airway obstruction will be determined
Symptoms of muscle weakness | 15 minutes after admission to the postanesthesia care unit
  The number of symptoms of muscle weakness measured 15 minutes after admission to the postanesthesia care unit will be determined

CONTACTS AND LOCATIONS:
Overall Officials: Glenn S Murphy, MD, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University HealthSystem, Evanston, Illinois, United States